CLINICAL TRIAL: NCT01384162
Title: An Open Label, Safety and Tolerability Continuation Study of Intracerebroventricular Administration of sNN0029 to Patients With Amyotrophic Lateral Sclerosis, Using an Implanted Catheter and SynchroMed® II Pump
Brief Title: An Open Label, Safety and Tolerability Continuation Study of Intracerebroventricular Administration of sNN0029 to Patients With Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Issues with development and supply of infusion system for delivery of IMP. Lack of favorable benefit risk ratio in sNN0029-003 study (review of interim data).
Sponsor: Newron Sweden AB (Industry)
Collaborators: Medtronic (Industry); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sNN0029-002
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; VEGF165; Safety; Intracerebroventricular; Infusion; Implantable
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sNN0029, ICV infusion (Experimental)
  Interventions: Drug: sNN0029

INTERVENTIONS:
Drug: sNN0029 — ICV infusion

SUMMARY:
This is an open label safety and tolerability continuation study of intracerebroventricular administration of sNN0029, containing the growth factor VEGF165, in patients with amyotrophic lateral sclerosis that have previously participated in study sNN0029-001. The intention of the study is to investigate safety and tolerability of intracerebroventricular administration of sNN0029 and whether it can improve motor function and prolong survival in patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ALS classified as definite, or probable with or without additional laboratory evidence, according to the revised WFN El Escorial criteria (Appendix B).
2. Previous participation in study sNN0029-001 with completion of 12 weeks study drug administration.
3. To have completed the investigations associated with safety in study sNN0029-001 without development of clinically significant safety concerns.
4. Patient has been given written and verbal information about the continuation study, has had the opportunity to ask questions about the study, and understands the time and procedural commitments.
5. Patient has given oral and / or signed consent (written) to participate in the study. In the event that a patient who gives oral informed consent is not physically able to sign the informed consent form (ICF) due to disease progression, a witness may sign the ICF on the patient's behalf.

Exclusion Criteria:

1. Hypertension defined as blood pressure >160 mmHg systolic or >90 mmHg diastolic.
2. Proliferative retinopathy.
3. Non-proliferative retinopathy of moderate severity or higher.
4. Concurrent clinically significant dementia as determined by the investigator.
5. Concurrent clinically significant depression as determined by the investigator.
6. Need for administration of any antiplatelet or anticoagulant medication (e.g. aspirin, Plavix, non-steroidal anti-inflammatory drugs [NSAIDs]). Low dose aspirin or occasional use of NSAIDs is allowed (See Appendix E).
7. Clinically significant abnormalities in haematology or clinical chemistry parameters as assessed by the investigator.
8. For female patients, ongoing pregnancy or planned pregnancy
9. Breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability through assessments of adverse events, vital signs, clinical laboratory tests, MRI of brain, fundus photography and device performance as characterized by catheter tip placement and infusion accuracy | multiple assessments over 120 weeks

SECONDARY OUTCOMES:
Disease activity as measured by ALS functional rating scale (FRS) - VEGF concentrations in CSF - Possible VEGF antibodies in plasma | Multiple assessments over 120 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wim Robberecht, MD, PhD, Principal Investigator — University Hospital Leuven, Department of Neurology
Locations (1):
- University Hospital Leuven, Department of Neurology, Leuven, Belgium